CLINICAL TRIAL: NCT01574547
Title: Risk Factors of Cat Scratch Colon Developing.
Acronym: CSC
Status: Completed | Type: Observational
Sponsor: University Hospital of the Nuestra Señora de Candelaria (Other)
Responsible Party: Principal Investigator, Juan-Salvador Baudet, Medical Doctor, University Hospital of the Nuestra Señora de Candelaria
Other Study IDs: Dig-3
Record Dates: First submitted 2012-04-08; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Mucosal Erosion
Keywords: Cat Scratch Colon.; Mucosal tears.; Mucosal erosion.; Colonoscopy.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cat Scratch Colon: Patients with mucosal tears during colonoscopy
- Control group: Patients without mucosal tears during the colonoscopy

SUMMARY:
This study was designed to: estimate the incidence of cat scratch colon in the investigators environment; explore the diseases associated to its development; identify the factors related to its development; and assess its clinical repercussions.

DETAILED DESCRIPTION:
All of the ambulatory colonoscopies performed at the investigators University Hospital from September 2007 were prospectively included in the study. Data recorded for each patient included: age, sex, disease background, reason for the examination, hematological data and the endoscopic diagnosis.

Every patient presenting CSC lesions had colon biopsies taken. These were studied by a single anatomic pathologist specializing in gastrointestinal pathologies.

The characteristics (age, sex, disease background, indication for surgery, age at the time of surgery, time elapsed since surgery, hematological data and pathoanatomical study of the colon biopsies) of diversion colitis patients with and without CSC lesions will bi compared.

ELIGIBILITY:
Inclusion Criteria:

* All of the ambulatory colonoscopies performed at our University Hospita

Exclusion Criteria:

* Patients thats refused.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All of the ambulatory colonoscopies performed at our Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10715 (Actual)
Dates: Start 2007-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Presence of cat scratch colon during the endoscopy | at the moment of colonoscopy
  Cat Scratch Colon: spontaneous tears appearing in the colon mucosa during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Juan-salvador Baudet, M.D., Principal Investigator — Ntra. Sra. de Candelaria University Hospital

REFERENCES:
- [Background] McDonnell WM, Loura F, Pointon MJ, Greenson JK. Cat scratch colon. Endoscopy. 2007 May;39(5):459-61. doi: 10.1055/s-2007-966266. PMID 17516354
- [Background] Cruz-Correa M, Milligan F, Giardiello FM, Bayless TM, Torbenson M, Yardley JH, Jackson FW, Wilson Jackson F. Collagenous colitis with mucosal tears on endoscopic insufflation: a unique presentation. Gut. 2002 Oct;51(4):600. doi: 10.1136/gut.51.4.600. No abstract available. PMID 12235088
- [Background] Yarze JC. Finding mucosal tears in collagenous colitis during colonoscopic insufflation. Gut. 2003 Apr;52(4):613-4; author reply 614. doi: 10.1136/gut.52.4.613-a. No abstract available. PMID 12631685
- [Background] Hata K, Watanabe T, Kanazawa T, Kazama S, Shida D, Nagawa H. Mucosal tears on endoscopic insufflation. Gut. 2003 Apr;52(4):613; author reply 613. doi: 10.1136/gut.52.4.613. No abstract available. PMID 12631686
- [Background] Mitchell JD, Teague R, Bolton R, Lowes J. Submucosal "dissection" in collagenous colitis. Gut. 2004 Mar;53(3):470. No abstract available. PMID 14960541
- [Background] Wickbom A, Lindqvist M, Bohr J, Ung KA, Bergman J, Eriksson S, Tysk C. Colonic mucosal tears in collagenous colitis. Scand J Gastroenterol. 2006 Jun;41(6):726-9. doi: 10.1080/00365520500453473. PMID 16716973
- [Background] Freeman HJ. Complications of collagenous colitis. World J Gastroenterol. 2008 Mar 21;14(11):1643-5. doi: 10.3748/wjg.14.1643. PMID 18350593
- [Background] van Velden R, Snieders I, Quispel R. Image of the month. Tearing of the colon in a patient with collagenous colitis during colonoscopy. Clin Gastroenterol Hepatol. 2010 Nov;8(11):A28. doi: 10.1016/j.cgh.2010.06.002. Epub 2010 Jun 25. No abstract available. PMID 20601144
- [Background] Baudet JS, Diaz-Bethencourt D, Arguinarena X, Soler M, Morales S, Aviles J. Cat scratch colon is caused by barotrauma secondary to insufflation during colonoscopy. Endoscopy. 2008 Oct;40(10):878; author reply 878-9. doi: 10.1055/s-2008-1077562. Epub 2008 Sep 30. No abstract available. PMID 18828090
- [Background] Baudet JS, Arguinarena X, Diaz-Bethencourt D, Soler M, Aviles J. [Cat scratch colon. A little known condition]. Rev Esp Enferm Dig. 2008 Dec;100(12):790-1. doi: 10.4321/s1130-01082008001200010. No abstract available. Spanish. PMID 19222340
- [Background] Purnak T, Ozaslan E, Yildiz A, Efe C. The cat scratch colon sign in a patient with chronic cholestasis. Endoscopy. 2010;42 Suppl 2:E117. doi: 10.1055/s-0029-1243983. Epub 2010 Mar 19. No abstract available. PMID 20306401
- [Background] Sherman A, Ackert JJ, Rajapaksa R, West AB, Oweity T. Fractured colon: an endoscopically distinctive lesion associated with colonic perforation following colonoscopy in patients with collagenous colitis. J Clin Gastroenterol. 2004 Apr;38(4):341-5. doi: 10.1097/00004836-200404000-00008. PMID 15087693